CLINICAL TRIAL: NCT00348699
Title: A Phase I Study and Pharmacological Trial of Once Weekly Aminoflavone Prodrug (AFP464) Administered 3 Out of Every 4 Weeks in Solid Tumor Patients
Brief Title: AFP464 in Treating Patients With Metastatic or Refractory Solid Tumors That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00164; NCI-2009-00164 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MAYO-IAB-05-00404800; MAYO-IAB-05-00404801; NCI-7380; CDR0000476275; MAYO-MC0513; MC0513 (Other: Mayo Clinic); 7380 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-12

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer; Recurrent Renal Cell Cancer; Stage IV Breast Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Primary Peritoneal Cavity Cancer; Stage IV Renal Cell Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Carcinoma, Ovarian Epithelial; Carcinoma, Renal Cell

ARMS (1):
- Treatment (AFP464) (Experimental): Patients receive AFP464 IV over 3 hours on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: AFP464; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: AFP464 — Given IV
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of AFP464 in treating patients with metastatic or refractory solid tumors that cannot be removed by surgery. Drugs used in chemotherapy, such as AFP464, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of AFP464 in patients with advanced solid tumors.

II. Evaluate the toxicity profile of AFP464. III. Characterize the plasma pharmacokinetics and urinary excretion of AFP464 and aminoflavone in these patients.

IV. Identify any activity of AFP464 in patients with metastatic cancer. V. Explore whether AFP464 induces cytochrome p450, family 1, member A1 (CYP1A1) expression in tumor (patients enrolled at the MTD) (patients enrolled at the MTD) and/or circulating tumor cells (CTCs) (dose-escalation phase and at the MTD).

VI. To explore the relationship between the pharmacogenetic analysis and toxicity or response.

OUTLINE: This is a dose-escalation study.

Patients receive AFP464 intravenously (IV) over 3 hours on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is now unresectable
* Patients with metastatic solid tumors who are refractory to available therapy or for whom standard systemic therapy does not exist
* Absolute neutrophil count (ANC) >= 1500/μL
* Platelets (PLT) >= 100,000/μL
* Total bilirubin =< upper limits of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine =< 1.25 x ULN; if above 1.25 x ULN calculated creatinine clearance must be >= 60 ml/min
* Hemoglobin (Hgb) >= 9.0 g/dl
* Normal diffusing capacity of the lung for carbon monoxide (DLCO) or the presence of an asymptomatic grade 1 DLCO; NOTE: DLCO must be corrected for hemoglobin
* Ability to provide informed consent
* Willingness to return to Mayo Clinic for follow-up
* Life expectancy >= 12 weeks
* Willingness to provide the biologic specimens (blood and urine) as required by the protocol
* COHORT II (MTD) PATIENTS ONLY:
* Patients with breast, ovarian, peritoneal or renal cell carcinoma
* Tumor that is amenable for biopsy taken during Cycle 1 at 24 +/- 4 hours following the end of AFP-464 infusion
* International normalized ratio (INR) =< 1.4
* Patients taking aspirin: discontinue >= 5 days prior to procedure
* Patients receiving IV Heparin: discontinue 4 hours prior to the procedure and an APTT measurement obtained if clinically indicated
* Patients receiving subcutaneous or low molecular weight heparin: discontinue for 8 hours prior to procedure

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 3 or 4
* Prior thoracic radiotherapy
* Symptomatic pulmonary disease
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, seizure disorder, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks prior to study entry
  * Mitomycin C/nitrosoureas =< 6 weeks prior to study entry
  * Immunotherapy =< 4 weeks prior to study entry
  * Biologic therapy =< 4 weeks prior to study entry
  * Radiation therapy =< 4 weeks prior to study entry
  * Radiation to > 25% of bone marrow
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* Uncontrolled brain metastases; Note: Brain metastases are not permitted on study unless the metastases have been treated by surgery or radiotherapy, and the patient has been neurologically stable and off steroids for >= 4 weeks
* Any of the following:

  * Pregnant women: Females of childbearing potential must have a negative serum pregnancy test =< 7 days prior to registration
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AFP464
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy
* Active smokers and those who have smoked =< 30 days prior to registration, and patients unwilling or unable to refrain completely from smoking while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-07; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, overall toxicity incidence, and toxicity profiles of AFP464 in the treatment of solid tumors | 28 days
  Measured by dose level and tumor site via the NCI CTCAE v 3.0. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Overall response of AFP464 in the treatment of solid tumors | Up to 3 months
  Measured by Modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Summarized by simple descriptive summary statistics delineating complete and partial responses as well as table and progressive disease in the two patient populations (overall and by tumor group).
Time to progression | From registration to documentation of progression, assessed up to 3 months
  Summarized descriptively.
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months
  Summarized descriptively.
Urinary excretion of AFP464 | Days 1-2, 8 and 15 of course 1
  Examined with descriptive summary statistics and simple graphical tools. Computed and correlated with toxicity and response via Spearman correlation coefficients for continuous variables or Wilcoxon rank sum test if one binary variable is involved.
Plasma area under the curve (AUC) of AFP464 | Days 1-2, 8 and 15 of course 1
  Examined with descriptive summary statistics and simple graphical tools. Computed and correlated with toxicity and response via Spearman correlation coefficients for continuous variables or Wilcoxon rank sum test if one binary variable is involved.

SECONDARY OUTCOMES:
Percent change in CYP1A1 | Baseline to 24 hours post AFP-464
  Computed and investigated with descriptive summary statistics and simple graphical tools. The percent change of CYP1A1 induction will also be correlated with response, toxicity, urinary excretion, and plasma pharmacokinetics measurements. circulating tumor cells (CTC) from all patients will be obtained pre- and post- infusion to determine the inducibility of gene expression of CYP1A1.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Goetz, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States